CLINICAL TRIAL: NCT06175325
Title: Pilot Study of the Safety and Efficacy of Trans-radial Superior Rectal Artery Embolisation for the Treatment of Haemorrhoids
Brief Title: Trans-radial Superior Rectal Artery Embolisation for Haemorrhoids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2602
Record Dates: First submitted 2023-11-21; First posted 2023-12-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhoids
Keywords: Embolisation
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-radial embolisation of haemorrhoids (Other): Haemorrhoids will be treated using arterial embolisation, using a trans-radial approach
  Interventions: Procedure: Trans-radial embolisation of haemorrhoids

INTERVENTIONS:
Procedure: Trans-radial embolisation of haemorrhoids — Once patients have provided informed consent to participate, an assessment of symptom severity will be obtained during the initial visit using the a standardised set of 4 validated scoring systems used in research of haemorrhoidal disease. These include the French bleeding score (FBS), Goligher classification of internal haemorrhoids (GS), quality of life score (QoL) and Visual analogue score for pain (VAS). Routine blood tests will be taken. During the procedure, routine observations will be recorded on the paper CRF. The data collected on the paper CRF will be entered onto the electronic CRF.
  The Transarterial fluoroscopically guided superior rectal artery embolization procedure will be performed on all participants. It is a day case procedure performed under local anaesthetic.

SUMMARY:
Endovascular embolisation is already a common procedure for bleeding haemorrhoids in the acute setting, where surgical options are not possible or have been exhausted. This pilot study aims to add to the small body of evidence that transarterial embolisation of symptomatic haemorrhoids is also safe and effective in the elective setting, providing a good alternative to conventional surgical management. This is a day case procedure that is performed under local anaesthetic. For selected patients, this presents a less invasive management option with reduced potential morbidity. For a health care system under significant financial stress, this provides a potential means of cost improvement, the extent of which this study will try and quantify. A series of 20 selected patients will be recruited to undergo this procedure and then followed up for 24 months. The long-term goal of this pilot study is to form the basis of a national registry of such procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the study must comply with all of the following prior to enrolment:

* Patients with grade II-IV haemorrhoid disease with re-current or active bleeding
* Patients with (i) who do not wish to undergo surgery for their symptoms
* Patients with (i) despite recent surgery
* Patients willing and able to give fully informed consent
* Patients aged ≥18 years

Exclusion Criteria:

* Patients who are not otherwise fit for surgery
* Patients with significant ano-rectal comorbidities (cancer, fistula, abscesses)
* Patient who are unable to sign the informed consent form.
* Patients who are pregnant (completed as part of standard IRMER protocol)
* Patients with history of significant colorectal disease or previous colectomy.
* Patients with history of an allergic reaction to x-ray contrast
* Patients who are currently involved in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and long-term effects | 3 years
  Safety and efficacy of the haemorrhoid embolisation procedure in relation to the rate of immediate and long-term complications

SECONDARY OUTCOMES:
Change of symptoms | 3 months
  Improvement in haemorrhoid related symptoms at 3 months using a questionnaire consisting of 4 standardised scoring systems. These include the French bleeding score (FBS), Goligher classification of internal haemorrhoids (GS), quality of life score (QoL) and Visual analogue score for pain (VAS).
Change of symptoms | 12 months
  Improvement in haemorrhoid related symptoms at 12 months using a questionnaire consisting of 4 standardised scoring systems. These include the French bleeding score (FBS), Goligher classification of internal haemorrhoids (GS), quality of life score (QoL) and Visual analogue score for pain (VAS).
Change of symptoms | 24 months
  Improvement in haemorrhoid related symptoms at 24 months using a questionnaire consisting of 4 standardised scoring systems. These include the French bleeding score (FBS), Goligher classification of internal haemorrhoids (GS), quality of life score (QoL) and Visual analogue score for pain (VAS).
Cost comparison | 3 years
  Comparison of the cost (in pounds £) associated with arterial embolisation, using a trans-radial approach to a traditional surgical operation
Procedural times comparison | 3 years
  Comparison with other similar studies using trans-femoral approach regarding procedural times
Radiation dose comparison | 3 years
  Comparison with other similar studies using trans-femoral approach regarding radiation dose
Contrast volume comparison | 3 years
  Comparison with other similar studies using trans-femoral approach regarding contrast volume

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No